CLINICAL TRIAL: NCT04720911
Title: Technology-Assisted Systems Change for Suicide Prevention
Acronym: TASCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Worcester Polytechnic Institute (Other)
Responsible Party: Principal Investigator, Celine Larkin, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H00020238; R34MH123578 (NIH)
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Suicide; Suicide, Attempted
MeSH Terms: conditions — Suicide; Suicide, Attempted | interventions — Aftercare

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-person TASCS (Experimental): This intervention is designed to assess the TASCS app administered via an in-person clinician in the ED, with follow-up telephone calls by a clinician
  Interventions: Behavioral: In-person TASCS; Behavioral: Follow-up care
- Telehealth TASCS (Active Comparator): This comparison condition is designed to assess the telehealth modality of TASCS in the ED (in contrast to in-person clinician modality), with follow-up telephone calls by a clinician
  Interventions: Behavioral: Telehealth TASCS; Behavioral: Follow-up care
- Self-administered TASCS (Active Comparator): This comparison condition is designed to assess the self-administered modality of TASCS (in contrast to clinician modality), with follow-up telephone calls by a clinician
  Interventions: Behavioral: Self-administered TASCS; Behavioral: Follow-up care

INTERVENTIONS:
Behavioral: In-person TASCS — In-person clinician delivery of the intervention, including the Safety Planning Intervention, connection to best-match behavioral health resources, and development of an outpatient treatment plan by a research clinician, facilitated by the TASCS Clinician App.
  Arms: In-person TASCS
Behavioral: Telehealth TASCS — Telehealth clinician delivery of the intervention, including the Safety Planning Intervention, connection to best-match behavioral health resources, and development of an outpatient treatment plan by a research clinician, facilitated by the TASCS Clinician App.
  Arms: Telehealth TASCS
Behavioral: Self-administered TASCS — Self-administration of the intervention, including the Safety Planning Intervention, facilitated by the TASCS ED Patient App.
  Arms: Self-administered TASCS
Behavioral: Follow-up care — Counseling calls and access to the Post-ED Patient and Family App for three months after the index presentation. These resources allow the patient and family to review their safety plan, life plan, and outpatient care plan

SUMMARY:
Effective prevention of suicide among adult emergency department (ED) patients hinges on an indispensable component: the ability to translate evidence-based interventions into routine clinical practice on a broad scale and with fidelity to the intervention components so they can have a maximum public health effect. However, there are critical barriers that prevent such translation, including a lack of trained clinicians, competing priorities in busy EDs, and incompatibility between requirements of evidence-based interventions (such as completing telephone coaching with patients after the ED visit) and the workflow and infrastructure typically present in most EDs. The proposed new intervention will address these barriers by building a suite of technologies that will make it easier to implement the Emergency Department Safety Assessment and Follow-up Evaluation (ED-SAFE), an evidence-based suicide intervention targeting perceived social support, behavioral activation and impulse control, revolutionizing the field's ability to scale and implement this intervention and acting as a model for efforts to implement other existing and emerging suicide interventions.

DETAILED DESCRIPTION:
The TASCS will be the first health information technology designed to enable flexible delivery of the ED-SAFE intervention components with strong fidelity and with responsiveness to the conditions and barriers present in most EDs. This will include an integrated approach to delivering components usually completed during the ED visit, such as personalized safety planning, as well as those completed after the visit, such as coaching to foster mental health treatment engagement. This R34 addresses both patient and implementation outcomes.

Aim 1 will use persona development, an innovative human computer interaction approach, to ensure the TASCS is intimately informed by end users.

Aim 2 will optimize the TASCS in a small field test in the ED.

Aim 3, modeled after a Hybrid Type 2 effectiveness-implementation design, will gather data on usability, acceptability, and implementation of the TASCS ED App using a randomized experiment (n=45) of three modalities: (1) On site (n=15), (2) Telehealth (n=15), and (3) Self-administered (n=15). For 3 months post-discharge, all participants will receive coaching calls, facilitated by the Post-ED Clinician App, and will have access to the Post-ED Patient and Family App. The intervention is intended to decrease suicidal ideation and behavior by improving perceived social support, increasing behavioral activation, and improving suicide-related impulse control.

Building a comprehensive suite of integrated enabling technologies to address ED-SAFE translation barriers will not only improve ED-SAFE intervention adoption, it will provide a road map for how to do the same for other suicide interventions, both existing and those yet to be developed, maximizing impact on the field.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Presenting to selected emergency departments during the study period
* Screened positive for active suicidal ideation in the past 2 weeks or attempt in the past 6 months
* Has a smartphone and access to the internet

Exclusion Criteria:

* Cognitively impaired (as assessed by study staff)
* <18 years of age
* Prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celine Larkin, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
NIMH will host the trial dataset on the National Database for Clinical Trials related to Mental Illness.

REFERENCES:
- [Derived] Larkin C, Tulu B, Djamasbi S, Garner R, Varzgani F, Siddique M, Pietro J, Boudreaux ED. Comparing the Acceptability and Quality of Intervention Modalities for Suicidality in the Emergency Department: Randomized Feasibility Trial. JMIR Ment Health. 2023 Oct 24;10:e49783. doi: 10.2196/49783. PMID 37874619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a large teaching hospital in the northeast United States, whose emergency department includes a dedicated psychiatric area. Recruitment took place at one emergency department at an academic medical center in the northeast U.S. between February 1 and September 15 2022.
Period: Overall Study
Arm/Group | In-person TASCS | Telehealth TASCS | Self-administered TASCS
Started | 15 | 16 | 16
Completed | 15 | 15 | 16
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: In-person TASCS: This intervention is designed to assess the TASCS app administered via an in-person clinician in the ED, with follow-up telephone calls by a clinician
- Active Comparator: Telehealth TASCS: This comparison condition is designed to assess the telehealth modality of TASCS in the ED (in contrast to in-person clinician modality), with follow-up telephone calls by a clinician
- Active Comparator: Self-administered TASCS: This comparison condition is designed to assess the self-administered modality of TASCS (in contrast to clinician modality), with follow-up telephone calls by a clinician
- Total: Total of all reporting groups
Arm/Group | Experimental: In-person TASCS | Active Comparator: Telehealth TASCS | Active Comparator: Self-administered TASCS | Total
Number analyzed (Participants) | 15 | 15 | 16 | 46
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [23 to 44] | 24 [21 to 33] | 27 [22 to 33] | 26.5 [22.75 to 37.50]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 7 | 6 | 10 | 23
  Male | 7 | 7 | 6 | 20
  Non-binary | 1 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 2 | 7
  Not Hispanic or Latino | 14 | 11 | 14 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 12 | 12 | 11 | 35
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1 | 2
Interpersonal Needs Questionnaire perceived burdensomeness subscale [Mean (Standard Deviation); unit: units on a scale] — Perceived burdensomeness as a subscale of the Interpersonal Needs Questionnaire (INQ-15). This subscale has a minimum score of 6 and maximum of 42, with a higher score representing higher perceived burdensomeness .
  units on a scale | 18.27 (10.47) | 20.67 (9.11) | 19.31 (11.06) | 19.41 (10.09)
Interpersonal Needs Questionnaire thwarted belongingness subscale [Mean (Standard Deviation); unit: units on a scale] — Thwarted belongingness as a subscale of the Interpersonal Needs Questionnaire (INQ-15; self-reported). This subscale has a minimum score of 9 and maximum of 63, with a higher score representing higher thwarted belongingness.
  units on a scale | 30.93 (15.43) | 38.60 (9.08) | 31.38 (13.88) | 33.59 (13.28)
Behavioral Inhibition & Activation Scales (BIS/BAS) Drive subscale [Mean (Standard Deviation); unit: units on a scale] — Behavioral activation as measured by the Drive subscale of the self-reported Behavioral Inhibition & Activation Scales (BIS/BAS). This Drive subscale has a minimum score of 4 and maximum of 16, with a higher score representing a better outcome.
  units on a scale | 10.33 (3.37) | 10.73 (3.01) | 12.38 (2.50) | 11.17 (3.04)
Suicide-related impulsivity [Mean (Standard Deviation); unit: units on a scale] — Suicide-related impulse control will be assessed the Recent Impulsivity Scale, a two-item scale ("How strong was the impulse (urgent need) to plan or to act in any suicidal way?"; "How difficult was it for you to suppress or to restrain the impulse to plan or to act in any suicidal way?") on a five-point scale from "Not at all" to "Extremely". The instrument has a minimum score of 1 and a maximum score of 5, with a higher score representing a worse outcome.
  units on a scale | 2.63 (1.27) | 3.10 (1.37) | 3.25 (1.44) | 3.00 (1.36)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Suicide Attempt in the Past Three Months
Description: Suicide Attempt is based upon participant response to "Actual Suicide Attempt" question within the "Suicidal and Self-Injury Behavior" subsection of the Columbia Suicide Severity Rating Scale (C-SSRS). The question is a yes/no with a "checking of the box" selection meaning yes, Actual Suicide Attempt and blank/unchecked means no, no Actual Suicide Attempt". We also reviewed the medical chart for ED presentations to ascertain whether the participant presented to the ED for a suicide attempt. The timeframe applied was past three months.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: In-person TASCS | Active Comparator: Telehealth TASCS | Active Comparator: Self-administered TASCS
Number analyzed (Participants) | 15 | 15 | 16
Participants | 0 | 1 | 1

2. Primary Outcome: Number of Patients With Active Ideation in Past Week at 3-month Follow-up
Description: Presence (yes/no) of active suicidal ideation within the past week as measured by the 'Suicidal Ideation (Most Severe)' subsection of the Columbia Suicide Severity Rating Scale.
Time Frame: 3 months
Population: Patients reachable by telephone at three months for follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: In-person TASCS | Active Comparator: Telehealth TASCS | Active Comparator: Self-administered TASCS
Number analyzed (Participants) | 7 | 10 | 10
Participants | 0 | 3 | 2

3. Secondary Outcome: Thwarted Belongingness From Interpersonal Needs Questionnaire (INQ-15)
Description: Thwarted belongingness as a subscale of the Interpersonal Needs Questionnaire (INQ-15). This subscale has a minimum score of 9 and maximum of 63, with a higher score representing higher thwarted belongingness.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: In-person TASCS | Active Comparator: Telehealth TASCS | Active Comparator: Self-administered TASCS
Number analyzed (Participants) | 7 | 10 | 10
units on a scale | 23.57 (4.08) | 26.70 (9.50) | 25.70 (12.39)

4. Secondary Outcome: Perceived Burdensomeness From Interpersonal Needs Questionnaire (INQ-15)
Description: Perceived burdensomeness as a subscale of the Interpersonal Needs Questionnaire (INQ-15). This subscale has a minimum score of 6 and maximum of 42, with a higher score representing higher perceived burdensomeness .
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: In-person TASCS | Active Comparator: Telehealth TASCS | Active Comparator: Self-administered TASCS
Number analyzed (Participants) | 7 | 10 | 10
units on a scale | 10.86 (4.91) | 11.30 (5.87) | 14.40 (11.05)

5. Secondary Outcome: Drive Subscale of the Behavioral Activation Scale (Continuous)
Description: Behavioral activation as measured by the Drive subscale of the Behavioral Activation Scale, part of the BIS/BAS Scale. This Drive subscale has a minimum score of 4 and maximum of 16, with a higher score representing a better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: In-person TASCS | Active Comparator: Telehealth TASCS | Active Comparator: Self-administered TASCS
Number analyzed (Participants) | 7 | 10 | 10
units on a scale | 11.43 (1.72) | 11.90 (1.85) | 12.20 (3.01)

6. Secondary Outcome: Suicide-related Impulse Control (Continuous)
Description: Suicide-related impulse control will be assessed the Recent Impulsivity Scale, a two-item scale ("How strong was the impulse (urgent need) to plan or to act in any suicidal way?"; "How difficult was it for you to suppress or to restrain the impulse to plan or to act in any suicidal way?") on a five-point scale from "Not at all" to "Extremely". The instrument has a minimum score of 1 and a maximum score of 5, with a higher score representing a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: In-person TASCS | Active Comparator: Telehealth TASCS | Active Comparator: Self-administered TASCS
Number analyzed (Participants) | 7 | 10 | 10
units on a scale | 1.29 (.39) | 1.40 (0.94) | 1.60 (0.99)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Death by suicide
Arm/Group | Experimental: In-person TASCS | Active Comparator: Telehealth TASCS | Active Comparator: Self-administered TASCS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT04720911/Prot_SAP_000.pdf